CLINICAL TRIAL: NCT00914602
Title: An Exploratory Pharmacokinetic, Pharmacodynamic and Safety Study of XP21279 (With Lodosyn®) and Sinemet® in Parkinson's Disease Subjects With Motor Fluctuations
Brief Title: An Exploratory Study of XP21279 (With Lodosyn®) and Sinemet® in Parkinson's Disease Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: XenoPort, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XP-C-058
Record Dates: First submitted 2009-06-03; First posted 2009-06-05 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination; Carbidopa

ARMS (2):
- Treatment Period A (Active Comparator): Treatment Period A: Sinemet® 25-100 treatment After screening all subjects will be placed on a fixed dosing Sinemet® time regimen for approximately 14 days.
  Interventions: Drug: Sinemet 25-100 Oral Tablet
- Treatment Period B (Experimental): Multiple-Dose XP21279 (with Lodosyn®) treatment. Upon completion of Sinemet® treatment eligible subjects will be placed on a fixed dosing time regimen of XP21279 (with Lodosyn®).
  Interventions: Drug: XP21279; Drug: Carbidopa Pill

INTERVENTIONS:
Drug: Sinemet 25-100 Oral Tablet — After screening all subjects will be placed on a fixed dosing Sinemet® time regimen for approximately 14 days.
  Other Names: Carbidopa / Levodopa
  Arms: Treatment Period A
Drug: XP21279 — Upon completion of Sinemet® treatment eligible subjects will be placed on a fixed dosing time regimen of XP21279 (with Lodosyn®).
  Other Names: XP21279 sustained related
  Arms: Treatment Period B
Drug: Carbidopa Pill
  Other Names: Lodosyn
  Arms: Treatment Period B

SUMMARY:
The purpose of the study is to assess the pharmacokinetics, pharmacodynamics, and safety of XP21279 sustained release formulation [administered with Lodosyn® (carbidopa)] and Sinemet® tablets in subjects with Parkinson's disease with Motor Fluctuations.

DETAILED DESCRIPTION:
This is a Phase 1/Phase 2 multiple-dose, multi-center, open-label, two period sequential-treatment study in subjects with Parkinson's disease to assess the pharmacokinetics, pharmacodynamics, and safety of XP21279 sustained release formulation [administered with Lodosyn® (carbidopa)] and Sinemet® tablets in subjects with Parkinson's disease and to explore dose correspondence between XP21279 and Sinemet® to guide dose selection for future studies in the target population (subjects with Parkinson's disease with motor fluctuations on Sinemet®).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with a clinical diagnosis of idiopathic Parkinson's disease, confirmed by the presence of at least two cardinal signs of the disease (resting tremor, bradykinesia, rigidity).
2. Subjects must have predictable motor fluctuations of the wearing off type, defined by wearing off in at least 50% of inter-dose intervals between the first and the last daily doses as recorded on the on/off diary over 3 days (Days -4 to -2) in the Screening Period.
3. Subjects must be on stable TID or QID Sinemet® or carbidopa/levodopa regimens from morning through early evening, with a total daily dose ranging from 400 mg to 1000 mg of levodopa, for at least 1 week prior to Screening.

Exclusion Criteria:

1. History, signs, or symptoms suggesting the diagnosis of secondary or atypical Parkinsonism.
2. Subject has greater than or equal to moderately disabling dyskinesias for greater than 25% of the waking day as assessed by a score of 2 or more on item 32 and a score of 2 or more on item 33 on the UPDRS at Screening.
3. Subjects who are dosing with Sinemet® or carbidopa/levodopa during the night time.
4. Subjects who have significant neurological symptoms not accounted for by Parkinson's disease.
5. Subjects who are taking concomitantly COMT inhibitors (i.e., entacapone or tolcapone) or treated with Stalevo®, Sinemet® CR, or Madopar®/Prolopa® (levodopa/benserazide).

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
to assess the pharmacokinetics of XP21279 sustained release formulation [administered with Lodosyn® (carbidopa)] and Sinemet® tablets in subjects with Parkinson's disease. | 4 weeks
  To establish a pharmacokinetic profile for XP21279
to assess the Pharmacodynamics of XP21279 sustained release formulation [administered with Lodosyn® (carbidopa)] and Sinemet® tablets in subjects with Parkinson's disease. | 4 weeks
  Changes in The Brief Parkinsonism Rating Scale during treatment
to assess the safety of XP21279 sustained release formulation [administered with Lodosyn® (carbidopa)] and Sinemet® tablets in subjects with Parkinson's disease. | 4 weeks
  Observe values and changes in clinical laboratory and vital sign parameters describe by time of collection for each treatment period.

SECONDARY OUTCOMES:
the dose correspondence between XP21279 and Sinemet® will be explored to guide dose selection for future studies in the target population | 4 weeks
  comparison of PK levels and doses.

CONTACTS AND LOCATIONS:
Overall Officials: Steve D Caras, MD, Study Chair — Arbor Pharma
Locations (2):
- United States (2):
  - XenoPort Investigational Site, Peoria, Arizona
  - XenoPort Investigational Site, Bingham Farms, Michigan